CLINICAL TRIAL: NCT00247364
Title: A Double Blind Crossover Trial of Levetiracetam (Keppra®) and Placebo in the Treatment of Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sleep Health Centers (Other)
Collaborators: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-P-001804
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2005-11-01 (Estimated); Status verified 2005-10

CONDITIONS: Restless Legs Syndrome
Keywords: RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam (Keppra)

SUMMARY:
To define the effective dose and tolerability of levetiracetam in individuals with Restless Legs Syndrome (RLS). It is hypothesized that levetiracetam will be well tolerated, safe and effective in treating the symptoms of RLS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic RLS according to the four IRLSSG diagnostic criteria

  1. An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs.
  2. The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as sitting or lying down.
  3. The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues
  4. The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night.

IRLS Rating Scale score greater than 15 at Baseline visit PLM-Index of 5 or greater during the first night of polysomnography Written informed consent obtained prior to any study procedures being performed.

Exclusion Criteria:

1. Women of childbearing potential, who have a positive urine pregnancy test or are lactating as the screening visit, or do not practice a clinically accepted method of contraception.
2. Individuals who are taking medication for Restless Legs Syndrome without a proper washout period
3. Individuals who are taking hypnotics, sedatives, antipsychotics, or neuroleptics
4. History of current diagnosis of other clinically relevant diseases that may confound assessments of RLS symptoms (e.g., Parkinson's disease, dementia, ALS, etc.)
5. Subjects with serum ferritin below 10µg/L
6. Subjects with an untreated sleep disorder that may confound assessments (e.g., narcolepsy, sleep apnea syndrome or other breathing-related sleep disorders, or REM sleep behaviour disorder)
7. Subjects with an apnea/hypopnea index of 15 or greater at the initial polysomnography visit
8. Subjects employed in shift work (e.g., employment hours disruptive to the normal circadian sleep-wake cycle such as nighttime or variable rotating shifts)
9. Subjects who have clinically significant or unstable medical conditions which in the opinion of the investigator would render the subject unsuitable for the study (e.g. severe cardiovascular disease, major depression, psychosis, hepatic or renal failure, etc.)
10. subjects with a positive urine drug test for illicit use of amphetamines, barbiturates, benzodiazepines, opiates, synthetic narcotics, and miscellaneous drugs commonly known as recreational drugs (e.g., cannabinoids including THC, heroine, cocaine)
11. Participation in any clinical drug or device trial in the 30 days prior to the screening visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-11; Study Completion 2005-10

PRIMARY OUTCOMES:
1:To investigate the efficacy of levetiracetam when used to treat RLS.
2:To assess tolerability and adverse event rates.

CONTACTS AND LOCATIONS:
Overall Officials: John W Winkelman, MD, PhD, Principal Investigator — Sleep Health Centers, Brigham and Women's Hosptial
Locations (1):
- Sleep Health Centers, Newton, Massachusetts, United States